CLINICAL TRIAL: NCT03113019
Title: Investigation of the Clinical and Laboratory Efficacy of Autogemotherapy Based on Autologous Antigen-activated Dendritic Cells in the Treatment of Patients With Breast Cancer
Brief Title: Autologous Antigen-activated Dendritic Cells in the Treatment of Patients With Breast Cancer
Acronym: BC-LDC
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Research Institute of Fundamental and Clinical Immunology (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Breast Cancer Lyzate DC
Record Dates: First submitted 2017-03-21; First posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-03

CONDITIONS: Breast Cancer
Keywords: dendritic cell, IL-12, IL-18, сytotoxicity
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients with breast cancer receive a cellular preparation consisting of dendritic cells loaded with tumor lysate antigens and activated mononuclear cells. Patients receive this treatment in the adjuvant mode at IIa-IIIc stages and in neoadjuvant regimen with progression or 4 stages of the disease
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Immunotherapy based on dendritic cells (Experimental): Intravenous administration dendritic cell and activated mononuclear cells at least 3 times 20-30 million cells / injection
  Interventions: Biological: Immunotherapy based on dendritic cells

INTERVENTIONS:
Biological: Immunotherapy based on dendritic cells — Intravenous injection of cells
  Other Names: Dendritic cell vaccine

SUMMARY:
The purpose of this work: to assess the tolerability and effectiveness of the autogemotherapy method on the basis of autologous antigen-activated dendritic cells in the treatment of patients with breast cancer.

This technology is intended for complex treatment of patients with breast cancer and is aimed at preventing the occurrence and treatment of secondary foci. The need for this technology is justified by the widespread occurrence of breast cancer among women, a decrease in the average age at onset of the disease and a young age, and the chemoresistantness of locally advanced forms of cancer.

DETAILED DESCRIPTION:
Currently, technologies are being developed to improve the clinical outcomes of patients with complex treatment of breast cancer. Many patients are immunosuppressed after surgical, radiation and chemotherapeutic treatment, which leads to dysfunction of T cells, resulting in tumor cells avoiding immune surveillance. Restoration of antitumor immunity during immunotherapy is one of the modern approaches in the treatment of breast cancer, which contributes to the formation of an effective specific immune response, the destruction of tumor cells while minimizing toxicity. Dendritic cells (DC) and the lymphocytes induced by them are one of the most effective methods for the destruction of residual cancer cells, which are the leading cause of relapse and metastasis.

ELIGIBILITY:
Inclusion Criteria:

1. For the first time established morphologically confirmed diagnosis of breast cancer
2. patients with II A, II B, IIIA, III B stages of breast cancer;
3. Patients with progressive or primary IV stage of breast cancer with cytologically confirmed and accessible soft tissue metastases;
4. Patients with HER-2 / neu 3 + positive and patients with triple negative breast cancer of the I-II stage (biologically unfavorable forms of breast cancer more prone to recurrence and metastasis).
5. Absence of severe somatic pathology in which medical intervention (at the stage of obtaining biological material or the stage of immunotherapy) will only worsen the patient's condition,
6. The patient's desire.

Exclusion Criteria:

1. Pregnancy at any time,
2. Impossibility of correction of therapy of concomitant diseases, if the taken preparations are proved to influence the immune status,
3. Rapid progression of the underlying disease, in which the use of immunotherapy is deontologically unjustified,
4. Individual intolerance to the components of the vaccine and / or the development of severe side effects on any of the components,
5. Refusal of the patient to participate in the study in oral or written form.
6. Patient involvement in any other clinical study (including those that the patient has not been informed by the direct oncologist who has been treated, but which has become known already after the beginning of any stage of the study).

Ages: 28 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-02-11 (Actual); Primary Completion 2017-02-11 (Actual); Study Completion 2017-09-11 (Estimated)

PRIMARY OUTCOMES:
Сytotoxicity | 6 months
  A study of the cytotoxic activity of peripheral blood mononuclear cells against tumor cells of the MCF-7 line. The result will be presented as the level of cytotoxicity (%) against the cells of the tumor line. The determination of cytotoxicity is carried out using a lactate dehydrogenase test (Promega). The level of the enzyme is proportional to the level of cytotoxicity.

SECONDARY OUTCOMES:
Parameters of peripheral blood | 6 months
  Leukocyte formula, the enzyme content (lactate dehydrogenase, alkaline phosphatase, liver enzymes) of C-reactive protein, creatinine
Immune status indicators | 6 months
  We investigated the content of CD 3, CD 4, CD 8, CD 19, CD 16, HLA-DR on CD 14 monocytes
The content of immunosuppressive populations | 6 months
  We investigated the content of T-regulatory cells, myeloid suppressors, myeloid and plasmacytoid dendritic cells
Interrogation of the patient using a visual analogue scale | 6 months
  patient evaluates his state in points. The patient is assessed such symptoms as fatigue, irritability, anorexia, nausea, pain, sleep disturbance)
Relapse-free period | 36 months
  A study of the period between the onset of complex treatment and immunotherapy until the recurrence of the disease.

CONTACTS AND LOCATIONS:
Overall Officials: Sergey V. Sennikov, MD, Study Director — RIFCI

IPD SHARING:
Plan to Share IPD: No